CLINICAL TRIAL: NCT02739529
Title: Dose-dense Paclitaxel (Genexol®-PM) Once a Week in Combination With Carboplatin Every 3 Weeks for Gynecologic Cancer (Adult Solid Tumor): a Phase I Trial
Brief Title: Study to Evaluate the Efficacy and Safety of Genexol-PM Once a Week for Gynecologic Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPMOC101
Record Dates: First submitted 2016-03-21; First posted 2016-04-15 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Gynecologic Cancer
MeSH Terms: interventions — genexol-PM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Genexol-PM 100mg/m2 IV infusion D1,D8,D15 Carboplatin 5 AUC IV infusion D1
  Interventions: Drug: Genexol-PM
- Cohort 2 (Experimental): Genexol-PM 120mg/m2 IV infusion D1,D8,D15 Carboplatin 5 AUC IV infusion D1
  Interventions: Drug: Genexol-PM
- Cohort 3 (Experimental): Genexol-PM 120mg/m2 IV infusion D1,D8,D15 Carboplatin 6 AUC IV infusion D1
  Interventions: Drug: Genexol-PM

INTERVENTIONS:
Drug: Genexol-PM — Cremophor EL-free polymeric micelle of paclitaxel

SUMMARY:
Dose-dense paclitaxel (Genexol®-PM) once a week in combination with carboplatin every 3 weeks for gynecologic cancer (adult solid tumor): a phase I trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who aged 20 years or older and under 80 year old female
2. Patients who were diagnosed histologically or cytologically or who were scheduled to reccur as an gynecologic cancer (epithelial ovarian cancer , fallopian tube cancer, primary peritoneal cancer, cervical cancer, uterine corpus cance, etc)
3. Patients seemed appropriate for Paclitaxel and Carboplatin combination therapy for the treatment
4. Patients whose ECOG performance score are 0-2
5. Patients who have adequate blood, kidney and liver function on screening within 14 days before the administration of the test drugs

   * Hb ≥ 10g/dl: Patients with less than 10g/dl of hemoglobin level were not allowed to use the test drugs unless they were recovered to 10g/dl or more.
   * ANC ≥ 1500/mm3
   * Platelet Count ≥ 100,000/mm3
   * Serum AST and ALT ≤ 2.5 X ULN
   * Serum ALP ≤ 2.5 X ULN
   * Serum creatinine ≤ 2.5 X ULN
6. Patients who participated voluntarily and who provided written informed consent before participating in the study

Exclusion Criteria:

1. Patients with the history of carcinoma in the past 5 years other than gynecologic cancer
2. Patients who received radiotherapy at abdominal cavity or pelvis
3. Patients who were receiving immunotherapy or hormone therapy
4. Patients who received a major surgery other than debulking surgery within 2 weeks before the screening
5. Patients with a past or present medical history of metastasis in central nervous system (CNS)
6. Patients with NCI CTCAE V4.0 Grade 1 or more sensory or motor neuropathy
7. Patients with severe comorbidities as follows

   * medical or mental condition impossible to understand the clinical trial and provide a written informed consent, based on the investigators' decision
   * severe cardiovascular disease (such as ischemic heart disease requiring medical therapy, myocardial infarction within the last 6 months, and grade 2~4 congestive heart failure defined by New York Heart Association criteria)
   * uncontrolled active infectious disease
   * hypersensitivity to the test drugs or the vehicle
8. Patients who participated in another study within 4 weeks before the screening
9. Pregnant, lactating women or Patients who do not use contraceptive methods that can be medically accepted to the possibility of pregnancy in female volunteers

Ages: 20 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) | 2 years
  MTD was determined as the dose where more than 2 out of 6 subjects experienced DLT
The recommended dose for the phase II study | 2 years
  Determined as the recommended dose for a phase 2 study based on the adverse events and toxicities at each dose groups

SECONDARY OUTCOMES:
The dose limiting toxicity (DLT) | 2 years
  Dose limiting toxicity (DLT) was defined as one of the following cases. NCI CTCAE V3.0 Grade 3 or more hypersensitivity despite premedication, Non-Hematological Toxicity other than nausea and vomiting, Hematological toxicity.
Toxicities | 2 years
  Clinical/laboratory toxicities were monitored after the treatment, in order to evaluate safety and tolerance of the test drugs, and adverse events, which were maintained until visit on discontinuation date, were followed until recovered or stabilized

CONTACTS AND LOCATIONS:
Overall Officials: Yong Man Kim, Principal Investigator — Asan Medical Center
Locations (1):
- Samyang Biopharmaceuticals, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No